CLINICAL TRIAL: NCT02359136
Title: Effect of Local Infiltration Anesthesia With Ropivacaine on Pain After Primary Total Hip Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 2012/1999
Record Dates: First submitted 2015-02-04; First posted 2015-02-09 (Estimated); Last update posted 2017-03-31 (Actual); Status verified 2017-03

CONDITIONS: Osteoarthritis, Hip
Keywords: Arthroplasty, Replacement, Hip; Anesthesia, Local; Ropivacaine; Randomized controlled trial
MeSH Terms: conditions — Osteoarthritis, Hip | interventions — Epinephrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LIA placebo (Placebo Comparator): local infiltration anesthesia using saline i addition to multimodal analgesic regimen
  Interventions: Procedure: local infiltration anesthesia using saline; Procedure: Multimodal analgesic regimen
- LIA Ropivacaine (Experimental): local infiltration anesthesia using Ropivacaine and Epinephrine i addition to multimodal analgesic regimen
  Interventions: Procedure: local infiltration anesthesia using Ropivacaine and Epinephrine; Procedure: Multimodal analgesic regimen

INTERVENTIONS:
Procedure: local infiltration anesthesia using Ropivacaine and Epinephrine — 150 ml Ropivacaine 2mg/ml + 0,5 ml Epinephrine 1 mg/ml: The first 50 ml will be injected in the periacetabular tissue after insertion of the acetabular component. After insertion of the femoral component, 50 ml will be inserted in the gluteus muscles and the proximal part of the iliotibial tract. The last 50 ml will be inserted in the subcutaneous layer.
  Arms: LIA Ropivacaine
Procedure: local infiltration anesthesia using saline — 150 ml 0,9% saline: The first 50 ml will be injected in the periacetabular tissue after insertion of the acetabular component. After insertion of the femoral component, 50 ml will be inserted in the gluteus muscles and the proximal part of the iliotibial tract. The last 50 ml will be inserted in the subcutaneous layer.
  Arms: LIA placebo
Procedure: Multimodal analgesic regimen — All patients will be operated under spinal anaesthesia with 2.0-3.0 ml Bupivacaine 0.5 % plain, preferably at the L2/L3 alternatively the L3/L4 vertebral interspace. Propofol infusion will be administrated for sedation if needed. Postoperative morphine will be given as needed intravenously when needed. After transfer to a specialized hip arthroplasty unit with a well-defined and experienced program for multimodal rehabilitation, multimodal oral opioid-sparing analgesia will be given to all patients; NSAIDS and Acetaminophen will be given at regular intervals and Oxycodone as needed.

SUMMARY:
Background: The Local infiltration analgesic (LIA) technique has been widely used to reduce opioid requirements and improve the patient's mobilization after total hip arthroplasty (THA). However, the evidence for LIA in THA remains to be clarified.

Purpose: To evaluate whether a single shot LIA in addition to a multimodal analgesic regimen reduces acute postoperative pain and opioid requirements after THA.

ELIGIBILITY:
Inclusion Criteria:

* all patients receiving total hip arthroplasty in the study period

Exclusion Criteria:

* contraindications to receive spinal anesthetic, Dexamethasone or Acetaminophen.
* Patients who received general anaesthetic
* patients who will get a different operation than standard direct lateral surgery
* Patients with osteosynthesis to be removed in the same operation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2014-03 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
postoperative pain assessed by numeric rating scale | 1 day (first postoperative day)
  assessed by numeric rating scale

CONTACTS AND LOCATIONS:
Overall Officials: Tina Strømdal Wik, md phd, Principal Investigator — St. Olavs Hospital
Locations (1):
- St.Olavs Hospital, Department of Orthopedics, Trondheim, Norway

REFERENCES:
- [Result] Hofstad JK, Winther SB, Rian T, Foss OA, Husby OS, Wik TS. Perioperative local infiltration anesthesia with ropivacaine has no effect on postoperative pain after total hip arthroplasty. Acta Orthop. 2015;86(6):654-8. doi: 10.3109/17453674.2015.1053775. Epub 2015 May 22. PMID 25997827